CLINICAL TRIAL: NCT04085627
Title: Comparative Open-label,Randomized, Fasting/Fed, Single Dose, Three-way Crossover Bioequivalence Study of Valsartan and Amlodipine Tablets (Hua Yuan Pharmaceutical LLC, China) and Valsartan and Amlodipine Tablets (Ⅰ) (Novartis Pharma Schweiz AG, Switzerland)
Brief Title: A Bioequivalence Study of Valsartan / Amlodipine From Valsartan and Amlodipine Tablets (Hua Yuan Pharmaceutical LLC, China) and Valsartan and Amlodipine Tablets (Ⅰ) (Novartis Pharma Schweiz AG, Switzerland)
Acronym: ABSVAFVATVAT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018-10-17
Record Dates: First submitted 2018-10-17; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Valsartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T Test (Experimental): Test drug(Valsartan / Amlodipine)1 tablet contains Valsartan 80mg& Amlodipine 5mg
  Interventions: Drug: Valsartan and Amlodipine Tablets
- R Reference (Active Comparator): Reference drug(Valsartan / Amlodipine)1 tablet contains Valsartan 80mg& Amlodipine 5mg
  Interventions: Drug: Valsartan and Amlodipine Tablets

INTERVENTIONS:
Drug: Valsartan and Amlodipine Tablets — 1 tablet contains Valsartan 80mg& Amlodipine 5mg

SUMMARY:
Comparative randomized, single dose, three periods, three-way crossover open-label study to determine the bioequivalence of Valsartan and Amlodipine Tablets (Hua yuan Pharmaceutical LLC, China) and Valsartan and Amlodipine Tablets (Ⅰ) (Novartis Pharma Schweiz AG, Switzerland).

DETAILED DESCRIPTION:
Primary Pharmacokinetic Parameters: Cmax, Area under cover (AUC0→t and AUC0→∞ ) .Secondary Pharmacokinetic Parameters: tmax and t1/2. The method of judging bioequivalence of three-cross-section repeating experiment design: first of all, the calculation of the SWR of the AUC and Cmax, if SWR≥0.294, the use of RSABE analysis; if Swr<0.294, the average Bioequivalence analysis method with Non-scale (bioequivalence limit is 80%~125 %）.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant non-lactating female, age 18 to 45 years, including the critical value.
* Male weight ≥ 50kg, female weight ≥ 45kg, body mass index (BMI) between 19 and 28kg / m2, including the critical value.
* Good health, no heart, liver, kidney, digestive tract, nervous system, mental disorders and metabolic disease history.
* Sign informed consent prior to the test and fully understand the contents, process and possible adverse reactions, and be able to communicate well with the researcher.

Exclusion Criteria:

* Any clinical trials in the 90 days prior to the trial, or other clinical trials planned for the duration of the trial.
* Underwent major surgery within 90 days of the trial or planned to undergo surgery within 3 months of the trial.
* Blood loss or blood donation over 300mL in the 90 days before the test.
* Esophageal reflux, stomach bleeding or peptic ulcer disease in the 180 days prior to the test, heartburn occurs more than once a week, or any surgical procedure that may affect drug absorption (E.G. cholecystectomy).
* Persons with specific allergies (asthma, urticaria, eczema, etc.) or allergies (such as those who are allergic to two or more medications, food or pollen), or are known to be allergic to the ingredients * or analogues of the drug.

  * The main components of the trial preparation: valsartan, benzene sulfonic acid amlodipine, microcrystalline cellulose, crosslinked povidone, crosslinked carboxymethyl cellulose sodium, silica, magnesium stearate, hydroxypropyl methyl cellulose, iron oxide yellow, polyethylene glycol, talc, Titanium dioxide; Reference Preparation main components: valsartan, amlodipine, microcrystalline cellulose, cross-linked povidone, silica, Magnesium stearate, hydroxypropyl methyl cellulose, iron oxide yellow, polyethylene glycol, talcum powder, Titanium Dioxide.
* Use of any medication within 28 days of the trial, including prescription, over- the-counter, and/or alternative medications (such as medicinal herbs, herbal medicines, hemostasis and blood-activating plants or health supplements), and the use of hormonal contraceptives or vaccines.
* A history of psychotropic substance abuse.
* Urine screening Positive.
* The average daily smoking was over 3 in the 90 days prior to the trial, alcohol consumption, women drinking more than 7 cups per week for 28 days or more than 14 cups per week for men (1 cups of =150ml wine =360ml Beer =45ml spirits).
* Alcohol expiratory test Positive.
* Body temperature (ear Temperature) ≥37.5℃, breathing is obviously abnormal and the researchers believe that it is not suitable to participate in the test, sitting systolic pressure >140mmhg or <100mmhg, sitting diastolic pressure >90mmhg or <60mmhg, sitting pulse 50 times/minute or > 100 Times/minute.
* Human immunodeficiency virus antibody (HIV-Ab), hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab) or Treponema pallidum antibody (TP) Positive.
* Special dietary requirements, No uniform diet during the trial.
* Subjects refused to comply with the drug before 48h banned caffeine, alcohol, grapefruit beverages and food (including tea, chocolate, coffee, coke, etc.).
* Participants with a companion refused to use effective contraceptive measures within 180 days of screening to the completion of the test, as detailed in Appendix 2.
* Female subjects were tested positive for blood/urine pregnancy.
* Persons with impaired renal function, or who have suffered from urinary system disease.
* A History of orthostatic hypotension.
* fainting during venipuncture, dizzy blood and venous blood collection difficult person.
* The physical examination was obviously abnormal and the researchers found it inappropriate to participate in the trial.
* There was a significant abnormality in the ECG test and the researchers found it inappropriate to Participate.
* Blood biochemistry, blood routine, urine routine examination had the obvious abnormality and the researcher thought that was not suitable to participate in the experiment.
* Subjects may not be able to complete this study or other researchers ' judgment for other reasons. Note: the exclusion criteria in 1th, 2, 3, 4, 6, 9 in the time are from the first 1 days before the administration of the Calculation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-12-26 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax | Up to 96 hours post dose in each treatment period
Bioequivalence based on AUC parameters | Up to 96 hours post dose in each treatment period

SECONDARY OUTCOMES:
Number of subjects with adverse events (AE)s | Up to 96 hours post dose in each treatment period
  Safety and tolerability parameters will include recording of AEs(blood biochemistry, urine routine examination, electrocardiograph, etc.)
blood pressure | Up to 96 hours post dose in each treatment period
  Vital sign measurement will include blood pressure
pulse rate | Up to 96 hours post dose in each treatment period
  Vital sign measurement will include pulse rate
respiration rate | Up to 96 hours post dose in each treatment period
  Vital sign measurement will include respiration rate
ear temperature | Up to 96 hours post dose in each treatment period
  Vital sign measurement will include ear temperature
complete blood count | Up to 96 hours post dose in each treatment period
  Clinical laboratory tests will include CBC

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Second Affiliated Hospital of WMU Phase I Clinical Trial Unit /Center Of Bioequivalence Study, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04085627/Prot_000.pdf